CLINICAL TRIAL: NCT06468397
Title: An Improved Retinal Detachment Repair Method: A First-in-human Clinical Trial of the Safety and Performance of the iSeelr™ Retinal Detachment Repair System to Seal Retinal Tears Intraoperatively
Brief Title: Acute Retinal Detachment Repair With the iSeelr™ Retinal Detachment Repair System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Photofuse Pty Ltd (Industry)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTF-CIP-01; CDMRP-W81XWH-21-1-0730 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs (CDMRP))
Record Dates: First submitted 2024-05-27; First posted 2024-06-21 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-08

CONDITIONS: Rhegmatogenous Retinal Detachment - Macula Off
Keywords: retinal detachment repair; laser; air; photocoagulation; photodehydration; gas tamponade; rhegmatogenous retinal detachment; 1940nm; retinal thermofusion; medical device; iSeelr™

STUDY DESIGN:
Intervention Model Description: First in human use of investigational device called iSeelr™ system for the treatment of Rhegmatogenous Retinal Detachment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Retinal Thermofusion (Experimental): Surgical treatment using the iSeelr™ medical device for retinal detachment repair
  Interventions: Device: iSeelr™

INTERVENTIONS:
Device: iSeelr™ — The iSeelr™ device will be used to deliver 1940nm laser output along with low airflow to seal a retinal tear

SUMMARY:
This study is a first-in-human clinical trial testing a new treatment for rhegmatogenous retinal detachments. The new treatment called retinal thermofusion uses a special laser device called iSeelr™ during surgery. The benefit of the device is that it repairs retinal tears without needing a gas bubble making it quicker to recover from surgery. The study will help us determine how safe and well the device performs in repairing a retinal detachment in people.

DETAILED DESCRIPTION:
The retina is a light-sensitive layer at the back of your eye that captures images. When light enters your eye, the retina turns it into signals that travel to your brain, helping you see. It's crucial for clear vision. When a retinal tear forms at the back of your eye, it can cause the fluid inside your eye to leak, leading to the retina peeling away and cause vision problems including blindness.

Retinal Thermofusion (RTF) uses a laser device called iSeelr™ to first dehydrate the fluid buildup around the retina and then laser treatment to seal the retina back in its place. The device was developed by Photofuse Pty Ltd and method validated in a laboratory with the Centre for Eye Research Australia and The University of Melbourne, Victoria, Australia.This clinical trial involves recruiting 10 participants with rhegmatogenous retinal detachment who will receive the treatment and be closely followed with 7 study visits over a three month period. This will allow us to assess the safety and performance of RTF. This research is being Sponsored by Photofuse Pty Ltd and is funded by the US Department of Defense (Award W81XWH-21-1-0730).

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or older.
* Willing and able to comply with all study requirements and visits.
* Provided written informed consent.

Study Eye:

* Recent onset as demonstrated by symptoms or diagnosis macular involving rhegmatogenous retinal detachment.
* Detachment due to single or multiple retinal tears in the superior region of the retina

Fellow eye:

• Visual acuity of 6/12 or better.

Exclusion Criteria:

* History of medical, surgical, or other conditions that, in the opinion of the investigator, would limit study participation e.g. unstable diabetes, poorly controlled hypertension.
* Travel limitations that could prevent review at proscribed study intervals or any other time during the study.
* Inability to provide informed consent.
* Anaesthetic risk factors or inability to lie supine for 1 hour.
* Pregnant and/or breast feeding (to be confirmed on treatment day)
* Current systemic infection
* Current ocular infection
* Unable to return for post-treatment visits
* Known inability to attend the emergency department in the event of an adverse event.

Exclusion criteria in the study eye:

* Significant vitreous haemorrhage partially or fully obscuring detailed examination of the retina
* Intraoperative identification of tears below the superior region in the area of retinal detachment not identified at the screening visit or during pre-operative examination. Note: Isolated retinal tears in attached retina, identified at any time are NOT an exclusion criterion and may be treated with lase as per standard of care
* Clinical signs of PVR (+1 flare, vitreous clumps, pigment clusters on the inferior retina, rolled retinal tear edge, star-fold)
* Myopia greater than -4 D spherical equivalent as confirmed by last refraction prior to becoming pseudophakic if cataract surgery has been performed
* History of glaucoma or elevated intraocular pressure >21mmHg
* Prior or current intraocular infection

Exclusion criteria in the fellow eye:

* Visual Acuity worse than 6/12
* Myopia greater than -4D spherical equivalent or axial length greater than 26mm if known
* Any potential sight threatening pathology in the fellow eye as determined by the investigator
* Extensive lattice degeneration
* Unilateral high myopia as determined by the investigator
* Family history of retinal detachment
* Collagen disorders such as Marfan's or Sticklers syndrome
* History of ocular trauma
* Evidence of any abnormality of the eye structure as determined by the investigator
* Planned surgery during the study period

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and performance of the investigational device, iSeelr™ System for the treatment of rhegmatogenous retinal detachments. | Assessment will take place before discharge on day of surgery and on days 1 and 2 post treatment
  Number of participants with successful retinal reattachment as defined by absence of leakage at the tear margin within the first 48 hours post-treatment without the need for gas tamponade
Assessment of intra-operative and post-operative adverse events | Up to 90 days post treatment
  To assess the safety of the treatment and the significance of any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Penelope Allen, FRANZO, Principal Investigator — The Royal Victorian Eye and Ear Hospital (RVEEH)
Locations (1):
- The Royal Victorian Eye and Ear Hospital (RVEEH), East Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed as a complete dataset in the Clinical Study Report

REFERENCES:
- [Background] Heriot WJ, Metha AB, He Z, Lim JKH, Hoang A, Nishimura T, Okada M, Bui BV. Optimizing Retinal Thermofusion in Retinal Detachment Repair: Achieving Instant Adhesion without Air Tamponade. Ophthalmol Sci. 2022 Jun 13;2(4):100179. doi: 10.1016/j.xops.2022.100179. eCollection 2022 Dec. PMID 36531586